CLINICAL TRIAL: NCT01777633
Title: Palliative Re-irradiation for Progressive Diffuse Intrinsic Pontine Glioma (DIPG) in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 027812-HMO-CTIL
Record Dates: First submitted 2013-01-13; First posted 2013-01-29 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2012-12

CONDITIONS: Pediatric Malignant Brain Tumor -Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- re-irradiation (Experimental): re-irradiation for progressive DIPG in children
  Interventions: Radiation: Palliative re-irradiation for progressive DIPG in children

INTERVENTIONS:
Radiation: Palliative re-irradiation for progressive DIPG in children

SUMMARY:
Although DIPG is not curable, re-irradiation with a modest total dose and short treatment time provides good palliation of symptoms, improves quality of life, delays disease progression and has minimal and manageable toxicity.

Treatment plan:

At progression, full radiological and clinical documentation necessary including a neurological exam by a neurologist will be done. Progressive patients will be referred to radiotherapy.

Radiation guidelines:

30.6 Gray (Gy) will be applied in 1.8 to 2Gy fractions in conformal radiation to tumor bed. Radiation will be done in standard accelerators and according to standard guidelines used in treatment for all brain tumor patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age:1 year-22 years
2. Patient/parent consent
3. Diagnosis of DIPG based on short classic history, clinical signs (long tract signs, cranial nerve deficits and ataxia) and classic MRI features (more than 2/3 of the tumor is located within the pons and tumor encompasses more than 60% of the pons)
4. A patient will be eligible for reirradiation if progression is diagnosed following a period of at least 4 months of stable disease after first irradiation.
5. Progression may be either clinical (new neurological deficit or worsening of an old deficit in two separate physical examinations) or radiological (tumor growth of >25%)

Exclusion Criteria:

1. Radiation necrosis post first irradiation
2. Unstable vital signs
3. Less than X months since previous irradiation

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
delaying disease progression | 1 year
  clinical progression: close follow up including biweekly neurological assessments to evaluate for clinical progression. any onset of a new neurological deficit or deterioration of an existing deficit will require follow up within one week. persistent deficit will be considered clinical progression.
  progression on imaging: MRI will be done every 3 months. tumor growth of >25% will be considered disease progression

SECONDARY OUTCOMES:
improving symptoms | 1 year
  parents will report daily ADL (Activities of Daily Living), brainstem functions including double vision, voice, swallowing functions and facial nerve palsy. parents will also report motor functions of the child in the biweekly visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel